CLINICAL TRIAL: NCT05341401
Title: Budesonide MMX Versus Prednisolone in Management of Mild to Moderate Ulcerative Colitis
Brief Title: Budesonide Multimatrix(MMX) Versus Prednisolone in Management of Mild to Moderate Ulcerative Colitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed Kamal Eldin Mohammed Ali, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Budesonide in UC
Record Dates: First submitted 2022-03-21; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Ulcerative Colitis Chronic
Keywords: ulcerative colitis.; Budesonide; prednisolone
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide MMX (Active Comparator): this study aims to detect the safety and side effects of budesonide MMX in the management of mild to moderate cases of ulcerative colitis in comparison to prednisolone. Budesonide MMX will be given after randomization to patients with mild to moderate cases who failed to respond to mesalazine. The dose will be 9mg as a single dose given for 8 weeks.
  Interventions: Drug: Budesonide MMX
- prednisolone (Active Comparator): this study aims to detect the safety and side effects of budesonide MMX in the management of mild to moderate cases of ulcerative colitis in comparison to prednisolone. prdinisolone MMX will be given after randomization to patients with mild to moderate cases who failed to respond to mesalazine. The starting dose will be 40 mg and reduced by 5 mg each weak for 8 weeks .
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Budesonide MMX — Budesonide MMX is a second generator corticosteroid with prolonged colonic release used for management of ulcerative colitis
  Arms: Budesonide MMX
Drug: Prednisolone — It is a corticosteroid used as a standard therapy for management of ulcerative colitis
  Arms: prednisolone

SUMMARY:
My study aims to directly compare the efficacy and safety of Budesonide MMX versus Prednisolone in the management of mild to moderate cases of ulcerative colitis.

DETAILED DESCRIPTION:
It is a randomized clinical trial where patients with mild to moderate ulcerative colitis who failed to respond to conventional therapy with mesalazine will randomly be divided into two groups one of them will be given prednisone and the other will be given budesonide MMX.

The efficacy of Budesonide MMX and Prednisolone will be measured by the rate of clinical, laboratory, endoscopic, and histological improvement 8 weeks after randomization. Clinical assessment (the rate of bowel movements and rectal bleeding) and laboratory investigations ( complete blood count [CBC], C reactive protein[CRP], and fecal calprotectin) will be done after 4 and 8 weeks from treatment initiation. Endoscopic and histological assessments will be done at week 8.

ELIGIBILITY:
Inclusion Criteria:

* This study will include patients with confirmed mild to moderate ulcerative colitis according to the Mayo score activity index with ages ranging between 18-60 years old.

Exclusion Criteria:

* Patients < 18 years old.

  * Pregnant females.
  * Patients with proven infection with any enteric pathogens (e.g., Shigella species, Clostridium species, Salmonella species, ova, parasites, Clostridium difficile toxins A or B, or HIV infection).
  * Patients who received oral or rectal steroids in the last 4 weeks, immunosuppressive agents in the last 8 weeks, or anti-tumor necrosis factor agents in the last 3 months.
  * Patients with severe colitis (Mayo score >11); Patients with evidence or history of toxic megacolon.
  * Severe anemia (hemoglobin <10.5 g/dl), leucopenia, or granulocytopenia.
  * Patients using any cytochrome P450 inducers or inhibitors (e.g., ketoconazole, phenytoin) or antibiotics.
  * Patients with renal disease/insufficiency.
  * Patients with type I diabetes.
  * Patients with glaucoma.
  * Patients with malignancies.
  * Patients with decompensated liver cirrhosis (Child-Pugh score B and C).
  * Patients with COVID 19 infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
comparison of the efficacy of both budesonide MMX and prednisolone. | 8 weeks
  To compare:
  - the clinical out come(by number of bowel movement, presence or absence of blood and abdominal pain) assessment will be done at 0 ,4 weeks and after 8 weeks from treatment initiation in both groups.
comparison of the efficacy of both budesonide MMX and prednisolone. | 8 weeks
  To compare:
  - laboratory out come ( CBC,CRP and fecal calprotectin) will be done at 0,4 and 8 weeks of treatment initiation
comparison of the efficacy of both budesonide MMX and prednisolone. | 8 weeks
  -to compare the : endoscopic out come using mayo scoring system.
comparison of the efficacy of both budesonide MMX and prednisolone. | 8 weeks
  to compare the histological remission

SECONDARY OUTCOMES:
incidence of side effects reported after using budesonide in mild to moderate cases of ulcerative colitis | 12 months
  to detect the side effects reported by the patients in each group and compare them to each other.
Types of side effects reported after using budesonide in mild to moderate cases of ulcerative colitis | 12 months

IPD SHARING:
Plan to Share IPD: Yes